CLINICAL TRIAL: NCT02242149
Title: Efficacy Study of Diacerein on Glycemic Control and Liver Fat in Type 2 Diabetes Subjects
Acronym: DGCLFT2DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Gil Fernando da Costa Mendes de Salles, PhD, Full Professor, Faculty of Medicine, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30194914.3.0000.5257
Record Dates: First submitted 2014-09-14; First posted 2014-09-16 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease
Keywords: Fat liver; Diabetes; Diacerein; Transient elastography; Treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Fatty Liver; Diabetes Mellitus | interventions — diacerein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): All subjects will be given placebo identically matched with regard to shape, color and taste. They will be given one tablet/day for 2 weeks and then two tablets/day for the duration of sudy.
  Interventions: Drug: Placebo
- Diacerein (Experimental): All subjects will be given diacerein with a starting dose of 50 mg in one tablet once daily for 2 weeks. After 2 weeks, they will be given diacerein 50 mg in one tablet twice daily for the duration of sudy.
  Interventions: Drug: Diacerein

INTERVENTIONS:
Drug: Diacerein — All subjects will be given diacerein with a starting dose of 50 mg in one tablet once daily for 2 weeks. After 2 weeks, they will be given diacerein 50 mg in one tablet twice daily for the duration of sudy.
  Other Names: Artrodar; Artifit; Acert
  Arms: Diacerein
Drug: Placebo — Sugar pill manufactured to mimic Diacerein
  Arms: Placebo

SUMMARY:
This study is conducted to test the hypothesis that in uncontrolled type 2 diabetic adults treatment with diacerein will improve glycemic control and will reduce liver fat within a 24 month period.

DETAILED DESCRIPTION:
Background: Recently, knowledge about diacerhein, an anthraquinone drug with powerful anti-inflammatory properties, revealed that this drug improves insulin sensitivity, mediated by the reversal of chronic subclinical inflammation. Amongst the numerous pathogenetic factors, oxidative stress and apoptosis of hepatocytes initiate many inflammatory processes and are involved in the progression of Non alcoholic fatty liver disease.

Aims:The aim is to evaluate the effect of treatment with diacerein in improvement of glycemic parameters (mean glycated hemoglobin, fasting blood sugar) and reduction of liver fat fraction.

Methods:Two-hundred patients will be randomly allocated either to treatment with diacerein plus their usual therapeutic regimen or to placebo for 24 months. Clinic, laboratory evaluation (including glycated hemoglobin, fasting blood sugar, creatinine, ferritin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), g-glutamyl transpeptidase, alkaline phosphatase, bilirubin, albumin, prothrombin time, platelet count, total cholesterol, high-density and low-density lipoprotein cholesterol and triglycerides and urinary albumin excretion rate no 24-hour urine collection) will be performed before and every 3 months until the end of study. Pro-Inflammatory cytokines, adiponectin and cytokeratin-18 were measured before, at 12 months and at the end of study. Liver fat fraction measurement using controlled attenuation parameter (CAP) by transient elastography. (Fibroscan) will be performed before and after the 12 and 24-month treatment, with the observers blinded to the allocation group.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes.
* Presence of liver steatosis diagnosed by ultrasound or transient elastography (Fibroscan®)
* Age 30-75 years.
* HbA1c 7.5- 9.5 for at least 8 weeks prior to screening.
* Stable diabetes therapeutic regimen consisting of either diet, oral hypoglycemic agents with or without insulin for 8 weeks prior to randomization.

Exclusion Criteria:

* Body mass index > 40 kg/m2
* Serum creatinine ≥180mmol/L or estimated glomerular filtration rate < 30 ml/min.
* Presence of any serious concomitant disease, such as a pulmonary disease or malignant disorders.
* Current daily alcohol ingestion ≥20 g.
* Hepatotoxic drugs.
* Presence of other chronic liver disease other than nonalcoholic fatty liver disease, including hepatitis B virus and hepatitis C virus infection, hemochromatosis, Wilson's disease, alfa-1 antitrypsin deficiency, autoimmune hepatitis.
* Women seeking pregnancy.
* Current use or previous use within 6 months of vitamin E or pioglitazone

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Evidence of improvement in glycemic control and improvement in liver steatosis | Within 12 and 24 months
  Reduction of mean glycated hemoglobin (≥ 1%) and reduction of liver fat fraction as measured by transient elastography (≥ 20%)

SECONDARY OUTCOMES:
Improvement of microalbuminuria | Within 24 months
  Reduction of albumin excretion rate on 24-hour urine collection
Changes of adipocytokines and cytokeratin-18 | Within 24 months
  Elevation of high molecular weight adiponectin and reduction of the apoptotic by-product cytokeratin (CK)-18

CONTACTS AND LOCATIONS:
Overall Officials: Gil F Salles, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Program of Arterial Hypertension, University Hospital Clementino Fraga Filho, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Cardoso CRL, Leite NC, Carlos FO, Loureiro AA, Viegas BB, Salles GF. Efficacy and Safety of Diacerein in Patients With Inadequately Controlled Type 2 Diabetes: A Randomized Controlled Trial. Diabetes Care. 2017 Oct;40(10):1356-1363. doi: 10.2337/dc17-0374. Epub 2017 Aug 17. PMID 28818994